CLINICAL TRIAL: NCT05940233
Title: Comparison of Rate of Complete Abortion Between Letrozole Plus Misoprostol vs Misoprostol Alone in First Trimester Pregnancy
Brief Title: Comparison of Rate of Complete Abortion Between Letrozole Plus Misoprostol vs Misoprostol Alone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 014/2566
Record Dates: First submitted 2023-05-24; First posted 2023-07-11 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Medical; Abortion, Fetus
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: We devide patient into 2 groups, intervention and control group. In intervention group we give the Letrozole 10 mg PO daily at day 1-3 prior to Misoprostol 800 mcg SL in day 4.
  In control group we give only Misoprostol 800 mcg SL.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole plus Misoprostol (Experimental): We give the Letrozole 10 mg PO daily at day 1-3 prior to Misoprostol 800 mcg SL in day 4.
  Interventions: Drug: Letrozole
- Misoprostol (Active Comparator): We give only Misoprostol 800 mcg SL.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — In the experimental group, we give the Letrozole 10 mg PO daily on the 4th day before Misoprostol 800 mcg SL on the 4th day. In the control group, we give Misoprostol 800 mcg SL on the 4th day.
  Other Names: Femara

SUMMARY:
Comparison of rate of complete abortion between Letrozole plus Misoprostol versus Misoprostol alone in first trimester pregnancy

DETAILED DESCRIPTION:
Comparison of rate of complete abortion between Letrozole plus Misoprostol versus Misoprostol alone in first trimester pregnancy; RCT

This reseach focus on the medical abortion in the early pregnancy loss. The target population is 70 patients (35 per group). We devide patient into 2 groups, intervention and control group. In intervention group we give the Letrozole 10 mg PO daily at day 1-3 prior to Misoprostol 800 mcg SL in day 4.

In control group we give only Misoprostol 800 mcg SL. Then, thepatien will follow up on day 7, TVS will be done to diagnose the complete abortion.

The primary outcome is rate of complete abortion between 2 groups. The secondary outcome is side effect of letrozole and induced to abortion time.

ELIGIBILITY:
Inclusion Criteria:

* Diafnoed Early pregnancy loss by TVS according to ACOG Practice bulletin 2018
* GA <= 14 weeks
* Os open <= 1 cm and no conceptus per os
* Hematicrit >= 30
* Systolic blood pressure >= 95 mmHg
* Informed consent done and can follow up and comunicate in Thai language

Exclusion Criteria:

* Allerguc to Letrozole or Misoprostol
* Intrauterine contraceptive device use
* Breast feeding
* Diagnoed with ectopic pregnancy or undiagnoed adnexal mass
* Severe or recurrent liver disease or AST or ALT more than or equal to 3 times of upper normal limit
* Multiple pregnancy
* Myoma uteri that involves the endometrium ex. Submucous myoma uteri
* Thromboembolism or has a history of thromboembolism
* Serum creatinine >= 2

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete abortion | up to 7 days
  Rate of complete abortion

SECONDARY OUTCOMES:
Side effect between both group | up to 7 days
  Number of patients with side effects between both group
induced to abortion time between both group | up to 6 months
  induced to abortion time between both group

CONTACTS AND LOCATIONS:
Overall Officials: ชื่นฤทัย ยี่เขียน, Ph.D., Study Chair — Queen Savang Vadhana Memorial Hospital, Thailand
Locations (1):
- Sutinee Srimahachota, Bangkok, Yannawa, Thailand

IPD SHARING:
Plan to Share IPD: No